CLINICAL TRIAL: NCT04125251
Title: Supporting Women and Girls in Pakistan: Scaling Up Empowerment and Care Strategies to Address Health and Survival
Brief Title: Men Engagement in Women Empowerment for Improving Maternal Mental Health Through Cash Transfer and Life Skills Building
Acronym: MEWE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Benazir Income Support Programme (BISP) (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OPP1148892
Record Dates: First submitted 2019-10-03; First posted 2019-10-14 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Empowerment; Domestic Violence; Depression; Self Efficacy
Keywords: Maternal Depression; Women Empowerment; Life Skills Building
MeSH Terms: conditions — Empowerment; Depression

STUDY DESIGN:
Intervention Model Description: The intervention and the assessment will be carried out parallel in the intervention and the control arm.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants, LSB providers and the outcomes assessors will not be having knowledge regarding the outcomes being assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BISP,CT & LSB to Couples (Active Comparator): In this arm 1, the LSB intervention will be offered to the BISP-CT beneficiary women and their spouses
  Interventions: Behavioral: Life Skills Building Training
- BISP,CT & LSB to Women (Active Comparator): In this arm, the LSB intervention will be offered to the BISP-CT beneficiary women only.
  Interventions: Behavioral: Life Skills Building Training
- BISP,CT & No LSB (No Intervention): This is the control group, where neither BISP-CT beneficiary women nor their spouses will be offered the LSB intervention

INTERVENTIONS:
Behavioral: Life Skills Building Training — The Life Skills Building intervention is a curriculum based on 10-12 sessions. The sessions will include the skills essential for family harmony and improving overall mental health of the participants
  Arms: BISP,CT & LSB to Couples; BISP,CT & LSB to Women

SUMMARY:
This project aims to offer Life Skills Building (LSB) intervention to Benazir Income Support Program (BISP) Cash Transfer (CT) beneficiaries in couples in order to reduce domestic violence and depression and improve women empowerment in married women of reproductive age. The intervention will be carried out in the rural settlements of district Thatta, Sindh Pakistan.

DETAILED DESCRIPTION:
The study will assess the impact of Life Skill Building (LSB) to Benazir Income support Program (BISP) Cash Transfer (CT) beneficiaries and their husbands in improving maternal mental and child health and its combined effect in empowering women and couples. The Formative phase of the project was dedicated for the development and modification of National level LSB curriculum for men and women. The formative phase was carried out in Thatta (Sindh), Rahimyar Khan (Punjab), Lasbela (Baluchistan) and Peshawar (KPK).

The intervention phase will be conducted in district Thatta, where BISP beneficiaries along with their spouses will be offered a LSB training. This intervention will be offered by community teachers to ensure sustainability and community trust. The participants will be recruited for baseline assessment followed by a comprehensive LSB intervention.The end-line follow up assessments (five months of intervention) will be done after the deliver of intervention. A qualitative summative inquiry will be done at the completion of the project to explore the overall impact of the LSB intervention. Since the project is being implemented with the BISP, the cost of intervention can be estimated for the scalability and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Adult married couples living together: where women receive Benazir Income Support Program (BISP) Cash Transfer (CT), have one child of at least 18 months and have no family migration plan for next 2 years

Exclusion Criteria:

* Gross mental impairment in either of the partners
* Either of the partner is physically challenged or bedridden

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The couples will be recruited from the list of adult women who are receiving Benazir Income Support Program (BISP) Cash Transfer (CT) and meet the eligibility criteria
Enrollment: 1696 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Decreased Maternal Depression | Base-line, and End-line (5 months post-intervention)
  The Patient Health Questionnaire (PHQ) is a self-administered instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day), over the last two weeks.
  PHQ-9 total score for the nine items ranges from 0 to 27. Scores of 5, 10, 15, and 20 represent cut points for mild, moderate, moderately severe and severe depression, respectively.
Decreased Domestic Violence | Base-line, and End-line (5 months post-intervention)
  The revised conflict tactics scale (CTS) consists of 20-item and is self-administered. The scale includes items regarding Negotiation (1-4), Psychological aggression (5-8), Physical assault (9-12), Sexual coercion (13-16) and Injury (17-20). The scoring criteria consists of a scale from 1-8, 1-6 indicates the frequency of conflict happened in the past year ranging from once to more than 20 times. 7 indicates conflict happened not in the past year but happened before that. If it never happened, 8 will be marked.
  There are many ways to score the CTS: Respondents who reported being a victim of or perpetrating an item or items (Prevalence). The number of times an item occurred in the past year (Frequency). Classifying each case into three categories: none, minor only, or severe (severity level). Classifying each case as respondent only, partner only, or both (mutuality types).
Improved General Self-Efficacy | Base-line, and End-line (5 months post-intervention)
  The General Self-Efficacy Scale (GSE) is a 10-item instrument to assess a general sense of perceived self-efficacy with the aim to predict coping and adaptation after stressful life events. Responses to each item are made on a 4-point scale: 1=Not at all true, 2=Hardly true, 3=moderately true, 4=exactly true.
  For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.

SECONDARY OUTCOMES:
Improved Household Food Security | Base-line, and End-line (5 months post-intervention)
  A six-item food security questionnaire (FSQ) is used to assess the food security in a household. The scale is valid, reliable and sensitive screening tool of food security in the household in the last 4 weeks, and whether the household was able to afford the food they needed.
  The total score ranges between 0-6, where score 0-1 shows high or marginal food security, score 2-4 shows low food security, score 5-6 shows very low food security.
Increased Resilience | Base-line, and End-line (5 months post-intervention)
  The validated Wagnild's resilience scale in Pakistani context will be used. The resilience scale comprise of five core characteristics of resilience that include: purposeful life, perseverance, equanimity, self-reliance and existential loneliness. It comprise of validated 14 items with 7-point Likert scale to rate the individual's evaluation ranging from 1 (Strongly Disagree) to 7 (Strongly Agree).
  Item scores are summed to yield a total score ranging from 14 to 98, with higher scores suggestive of greater perceived resilience categorized as very low (14-56), low (57-64), on the low end (65-73), moderate (74-81), moderately high (82-90), and high (91-98).
Improved Gender Attitude | Base-line, and End-line (5 months post-intervention)
  The Gender Equitable Attitude Scale (GEAS) is a 21 item Likert scale ranging from 4 (strongly agree) to 1 (strongly disagree). It has been adapted from 34-item original "The Gender-Equitable Men Scale (GEM Scale)" and 13-item "Gender Equitable Men Scale" adapted in the context of Pakistan. The total score ranges from 21-84, where higher score shows more gender equitable attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar ZB Bhutta, PhD, Principal Investigator — The Aga Khan University, Karachi, Pakistan; Rozina RK Karmaliani, PhD, Study Director — The Aga Khan University, Karachi, Pakistan; tazeen TS Ali, PhD, Study Director — The Aga Khan University, Karachi, Pakistan
Locations (1):
- The Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The IPD will be analyzed using unique identifiers and only the study results will be shared through publications

DOCUMENTS (2):
  • Study Protocol (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT04125251/Prot_003.pdf
  • Informed Consent Form (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT04125251/ICF_004.pdf